CLINICAL TRIAL: NCT03281785
Title: Ultrasound Evaluation of the Diaphragmatic Musculature in Mechanically Ventilated Patients in Intensive Care Unit
Brief Title: Ultrasound of Diaphragmatic Musculature in Mechanically Ventilated Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: MD%2f16.12.52
Record Dates: First submitted 2017-09-11; First posted 2017-09-13 (Actual); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Mechanical Ventilation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pressure controlled mandatory ventilation mode (P-CMV) (Active Comparator): Patients will be ventilated using pressure controlled mandatory ventilation mode
  Interventions: Other: Pressure controlled mandatory ventilation mode (P-CMV)
- Pressure synchronized intermittent mandatory ventilation (Active Comparator): Patients will be ventilated using pressure synchronized intermittent mandatory ventilation mode (P-SIMV)
  Interventions: Other: Pressure synchronized intermittent mandatory ventilation
- Pressure support mode (PS) (Active Comparator): Patents will be ventilated with pressure support mode (PS)
  Interventions: Other: Pressure support mode (PS)

INTERVENTIONS:
Other: Pressure controlled mandatory ventilation mode (P-CMV) — Pressure controlled mandatory ventilation mode (P-CMV)
  Arms: Pressure controlled mandatory ventilation mode (P-CMV)
Other: Pressure synchronized intermittent mandatory ventilation — Pressure synchronized intermittent mandatory ventilation
  Arms: Pressure synchronized intermittent mandatory ventilation
Other: Pressure support mode (PS) — Pressure support mode (PS)
  Arms: Pressure support mode (PS)

SUMMARY:
Muscle weakness and dysfunction are common problems in patients hospitalized in the intensive care unit. Respiratory muscle weakness during mechanical ventilation was recognized a state of muscular fatigue. The terminology 'ventilator-induced diaphragmatic dysfunction' (VIDD) originally was introduced to describe these effects of mechanical ventilation and respiratory muscle unloading on the diaphragm.

Ultrasonography is becoming increasingly popular management of ICU patients. It is a simple, non-invasive and safe imaging technique that can be used for the assessment of distinctive diaphragmatic characteristics.

Parameters such as amplitude and velocity of contraction, which can be assessed using M-mode ultrasound. In addition, static and dynamic (thickening fraction during inspiration) diaphragmatic thickness can also be measured by ultrasonography.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the effect of different modes of mechanical ventilation on diaphragmatic thickness using ultrasonography and the relation between time of mechanical ventilation and the percentage of change of diaphragmatic thickness in head trauma patients subjected for mechanical ventilation (>2 days) intensive care unit.

Modes of ventilation will be used in the study are:

* Pressure controlled mandatory ventilation mode (P-CMV).
* Pressure synchronized intermittent mandatory ventilation mode (P-SIMV).
* Pressure support (PS) mode.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status grades I and II.
* Glasgow coma scale < 8.
* Selections of patients need mechanical ventilation (>2 days).
* Head trauma patients.

Exclusion Criteria:

* History of diaphragmatic disease
* Neuromuscular disease
* Anatomical malformation of the diaphragm.
* Patients with chest disease
* Diabetic patients.
* Chest trauma
* Chest malignancy.
* Use of non-invasive ventilation before the start of invasive ventilation.
* Selection of patients of short period of mechanical ventilation (< 2 days).
* Hemodynamic instability.
* Morbid obesity (body mass index > 40 kg/m2).

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 93 (Actual)
Dates: Start 2017-09-20 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Diaphragmatic thickness | for 3 weeks after initiation of mechanical ventilation
  changes in diaphragmatic thickness from baseline to nadir

SECONDARY OUTCOMES:
The relation between time of mechanical ventilation and the percentage of change of diaphragmatic thickness | for 3 weeks after initiation of mechanical ventilation
  measurement of the diaphragmatic thickness as usual and calculate the percentage of change of the diaphragmatic thickness over the time of mechanical ventilation
Glasgow coma scale (GCS) | for 2 weeks after initiation of mechanical ventilation.
Sequential organ failure assessment (SOFA) score | for 3 weeks after admission to the ICU
Complete blood picture | for 3 weeks after admission to the ICU
Coagulation profile | for 3 weeks after admission to the ICU
Liver function | for 3 weeks after admission to the ICU
Renal function tests | for 3 weeks after admission to the ICU
Mean blood pressure | for 3 weeks after admission to the ICU
Heart rate | for 3 weeks after admission to the ICU
Arterial Oxygen Saturation | for 3 weeks after admission to the ICU
Central Venous Pressure | for 3 weeks after admission to the ICU
temperature | for 3 weeks after admission to the ICU
mode of ventilation | for 3 weeks after initiation of mechanical ventilation
tidal volume | for 3 weeks after initiation of mechanical ventilation
respiratory rate | for 3 weeks after initiation of mechanical ventilation
airway pressure | for 3 weeks after initiation of mechanical ventilation
  peak and mean airway pressure
ICU stay | for 3 weeks after initiation of mechanical ventilation
  Time from admission to the ICU untill discharge or death
Duration of mechanical ventilation | for 3 weeks after initiation of mechanical ventilation
  time from initiation of mechanical ventilation till extubation or death

CONTACTS AND LOCATIONS:
Overall Officials: Amal R Ali, MD, Study Chair — Professor of Anesthesia and Surgical Intensive Care; Hanaa M Elbendary, MD, Study Director — Professor of Anesthesia and Surgical Intensive Care
Locations (1):
- Mansoura University, Faculty of Medicine, Al Mansurah, DK, Egypt

IPD SHARING:
Plan to Share IPD: Undecided